CLINICAL TRIAL: NCT05434026
Title: Chinese Colorectal Cancer Database
Acronym: CCCD
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Peking University People's Hospital (Other); Peking University Cancer Hospital & Institute (Other); Peking Union Medical College Hospital (Other); The First Hospital of Jilin University (Other); Ruijin Hospital (Other); First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, Director of general surgery, principal investigato, Beijing Friendship Hospital
Other Study IDs: CCCD
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Colonic Cancer; Rectal Cancer; Prospective Studies
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To establish the Chinese people's own clinical data database of colorectal cancer, reflecting the law and characteristics of colorectal cancer patients in China.
2. Based on colorectal cancer surgery, collect clinical data, especially data on clinical manifestations, complications, laboratory tests, auxiliary examinations, postoperative clinical effects, surgical complications, and colorectal cancer recurrence, so as to lead the direction of clinical practice and academic research of colorectal cancer surgery in China. It provides a certain basis for future research on colorectal cancer.
3. Provide academic consultation and data support to national health authorities.

ELIGIBILITY:
Inclusion Criteria:

* adenocarcinoma of the colon by biopsy
* tolerable to surgery
* be able to understand and willing to participate in this trial with signature

Exclusion Criteria:

* can not tolerate the surgery
* history of serious mental illness
* the researchers believe the patients should not enrolled in

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: colorectal cancer patients who are suitable and willing to accept the surgery and also agree with the trial
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2022-08-03 (Estimated); Primary Completion 2032-06-22 (Estimated); Study Completion 2032-06-22 (Estimated)

PRIMARY OUTCOMES:
Positive rate of circumferential resection margin (CRM) of the specimens | 10 days after surgery
  Circumferential resection margin (CRM) is the distance between the deepest point of tumor in the primary cancer and the margin of resection in the retroperitoneum or mesentery by pathological examination. CRM 0-1mm is defined as positive, while >1mm is negative.
The grade score of the specimens integrity | 10 days after surgery
  shows the quality of the specimens: grade 1 is bad gross specimen which means incomplete mesorectum and pelvic fascia, and muscle layer can be see >5mm; grade 3 is high quality gross specimen, which means the specimen is cylindrical, mesorectum and pelvic fascia are complete; grade 2 is between 1and 3.
The distance between lower tumor margin and the lower reaction margin | 10 days after surgery
  shows the oncological safety of the surgery by pathological examination. Reports should contain the distance between lower tumor margin and the lower reaction margin.
local recurrence rate | 3 years after surgery
  show the oncological efficacy by 3-year follow-up according to the NCCN guideline. Participants should report every follow-up examinations which prove tumor recurrence and/or metastasis or not.
the operative time | 30 days after surgery
  preoperative safety containing operation information, complication information.
postoperative hospital stay | 3 year after surgery
  recovery information.
the score of postoperative life | 6 months after surgery
  quality of life contains two scales: Wexner scale and EORTC QLQ-CR29 scale, which show quality of life and the anal function.
disease free survival rate | 3-year after surgery
  show the oncological efficacy by 3-year follow-up according to the NCCN guideline. Participants should report every follow-up examinations which prove tumor recurrence and/or metastasis or not.
overall survival rate | 3-year after surgery
  show the oncological efficacy by 3-year follow-up according to the NCCN guideline. Participants should report every follow-up examinations which prove tumor recurrence and/or metastasis or not.
the rate of postoperative complications | 30 days after surgery
  preoperative safety containing operation information, complication information.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongtao Zhang, Beijing, China